CLINICAL TRIAL: NCT02196987
Title: Pain Level During Male Urethral Catheterisation - Does Patient Attempted Urination During Catheterisation Reduce Pain? A Prospective Randomized Study
Brief Title: Does the Act of Urination During Urethral Catheterisation in Males Reduce Pain?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Kobi Stav, Assaf-Harofeh Medical Center
Other Study IDs: 109/14
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Pain
Keywords: Pain; Catheter; Urethra; Urination
MeSH Terms: conditions — Pain | interventions — Urinary Catheterization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Urination, urethral catheterisation: Act of urination during urethral catheterisation in males
  Interventions: Other: Urination during urethral catheterisation
- Lie, catheterisation, urethra: Urethral catheterisation without medical professional guidance
  Interventions: Other: Urethral catheterisation, without further guidance

INTERVENTIONS:
Other: Urination during urethral catheterisation — Requesting the patient to urinate while inserting urethral catheter
  Groups: Urination, urethral catheterisation
Other: Urethral catheterisation, without further guidance — Lying, inserting urethral catheter, without further guidance from health care professional
  Groups: Lie, catheterisation, urethra

SUMMARY:
Currently, there are no specific guidelines or best practice suggestions for best male catheterization as fat as insertion technique. There is however, information as to reducing infection, and as to recommended lubricant.

From our experience, the investigators have noticed that when requesting the patient to attempt urination while inserting a urethral catheter, the level of pain and discomfort is reduced. In this study, the investigators will evaluate the pain level during male urethral catheterization in each technique.

Our hypothesis is that the level of pain will be much less if the in the study group where the act of urination will be requested from the patient.

DETAILED DESCRIPTION:
This is a randomized prospective study that will compare the pain levels of urethral catheterization in men randomized to requesting to urinate while inserting a urethral catheter to normal catheter insertion.

Males aged 18 years and older who will be referred for multichannel Urodynamic study in order to evaluate lower urinary tract symptoms will be included.

Patients will be randomized to 2 groups: (1) Patients who will be requested to urinate while catheterising the urethra to its full length; (2), Patients who will be requested to lie while catheterising the urethra, without further instructions from the medical professional. In both groups, prior to catheterisation, 10 ml of lidocaine gel will be inserted into the urethra. The randomization technique will be employed by a computerized random number generator.

A 12F Tieman urethral catheter will be introduced in order to measure post-void residual volumes. Subsequently, multichannel Urodynamic testing (Duet Encompass System - Mediwatch Group Plc) will be performed using a dual lumen 6F urethral and 9F rectal catheters. Filling will be carried out using room temperature saline at a filling rate of 50 ml/min.

Patients will be requested to fill out a 0 (no pain) to 10 (worst imaginable pain) visual analog pain scale (VAS) in different time points: before the procedure (baseline), immediately after gel instillation, immediately after the introduction of the Tieman catheter, 15 minutes after the catheter will be taken out.

Time frame of the study: 30 minutes before the test and 1 hour after the test. Since the study evaluates pain during the procedure the time frame of the study and assessment is very short. longer follow-up is not needed.

ELIGIBILITY:
Inclusion Criteria:

* men aged 18 years and older who will be referred for multichannel Urodynamic study in order to evaluate lower urinary tract symptoms.

Exclusion Criteria:

* use of any analgesics within the previous 24 hours, known urethral stricture, active urinary tract infection, indwelling urethral catheter, pre-existing urethral pain (e.g. patients with chronic pelvic pain syndromes and interstitial cystitis), inability to cooperate with pain assessment due to mental disorders.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men who will be referred to Urodynamic study
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in visual analog pain scales | Before catheterisation, during catheterisation, 15 minutes after catheterisation
  A 0 to 10 visual analog pain scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Kobi Stav, MD, Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Beer Yaakov, Zeriffin, Israel